CLINICAL TRIAL: NCT04188314
Title: A Randomised Control Trial to Compare Quality of Recovery Between Desflurane and Isoflurane Inhalational Anaesthesia in Patients Receiving General Anaesthesia for Ophthalmological Surgery at Dr. George Mukhari Academic Hospital
Brief Title: Comparing Quality of Recovery Between Desflurane & Isoflurane in Eye Surgery Patients at Dr George Mukhari Acad Hospital
Acronym: DIQoR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sefako Makgatho Health Sciences University (Other)
Responsible Party: Principal Investigator, Dr. Charle Steyl, Registrar in Department of Anaesthesiology, Sefako Makgatho Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMUREC/M/240/2019:PG
Record Dates: First submitted 2019-10-27; First posted 2019-12-05 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Quality of Recovery; Anesthesia Recovery Period
Keywords: Anesthesia: General; Outcome; Quality of Recovery Score; Anesthetics: Volatile; Desflurane; Isoflurane
MeSH Terms: interventions — Desflurane; Isoflurane

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomised, controlled, patient and observer blinded, single-centre trial with two parallel groups and a primary end-point of 15-point Quality of Recovery Score on day 1 after surgery. Randomization will be performed as block randomization with a 1:1 allocation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded (masked) to the group they have been randomised to, as the vapour will only be started after induction of anaesthesia. The research assistant administering the post-operative QoR-15 will be blinded (masked) to the intervention.
  The treating anaesthetist, the Chief Researcher and theatre staff will not be blinded to the intervention, as this would not be practical. All treating anaesthetists and theatre staff will be strongly inculcated not to disclose the allocation status of the participant at any time prior or after the general anaesthetic.
  The piece of paper indicating the group will be attached to the Case Report Form. The Case Report Form will be collected by the Chief Researcher and will not be in the patient's file where it may unblind the patient or research assistant.
  There are no circumstances under which unblinding will be permissible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane Interventional Group (Experimental): The intervention group will receive desflurane for maintenance of anaesthesia. Standard protocols for induction and maintenance of anaesthesia will be followed, as discussed with Prof. F. Puehringer, an international expert in the field of desflurane use. A detailed leaflet describing the protocol has been developed, which will be handed to the treating anaesthetist on the day of surgery.
  After induction of anaesthesia and after the airway is secured, fresh gas flow is reduced to 2 l/min and the desflurane vaporiser is opened to 12%. This is maintained until 1MAC is reached. The fresh gas flow will then be turned down to 0.2-0.5 l/min (taking into consideration the machine leak) and the vaporiser adjusted to maintain 1MAC. The use of basal to minimal fresh gas flow is intentional, to minimise the amount of anaesthetic vapour used. When basal flow is used, 100% oxygen is required to meet oxygen demand.
  Interventions: Drug: Desflurane
- Isoflurane Control Group (Active Comparator): The control group will receive Isoflurane for maintenance of anesthesia. After induction of anaesthesia and after the airway is secured, fresh gas flow is reduced to 2 l/min and the Isoflurane vaporiser is opened and adjusted to attain 1MAC. Once 1MAC is attained, the fresh gas flow will be reduced to 0.2-0.5 l/min (taking into consideration the machine leak) and the vaporiser will be adjusted to maintain 1MAC. The use of basal to minimal fresh gas flow is intentional, to minimise the amount of anaesthetic vapour used. When basal flow is used, 100% oxygen is required to meet oxygen demand.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Desflurane — The intervention group will receive desflurane for maintenance of anaesthesia, and the quality of recovery score will be compared post-operatively with the control group who received isoflurane.
  Other Names: Suprane
  Arms: Desflurane Interventional Group
Drug: Isoflurane — The control group will receive Isoflurane for maintenance of anesthesia. The quality of recovery score will be compared post-operatively with patients in the intervention group who received desflurane.
  Other Names: Forane
  Arms: Isoflurane Control Group

SUMMARY:
Recovery after surgery and anaesthesia has traditionally been assessed with objective measures including time to awakening, time to regaining airway reflexes, duration of stay in the recovery room and/or hospital, and incidence of adverse events like pain and post-operative nausea and vomiting.

Increasingly, the patient's experience of their post-operative recovery is being recognised as an important outcome after surgery. The 15-Item Quality of Recovery score (QoR-15) has been validated to give a patient-centred global measure of overall health status after surgery and anaesthesia. This score has recently been translated and validated in isiZulu.

Desflurane is the newest anaesthetic vapour to market, with many benefits from the anaesthetist's perspective: faster time to awakening, faster time to regaining airway reflexes, and a clearer sensorium post-operatively. However, there is a paucity of data evaluating whether this translates to better quality of recovery for the patient. Desflurane is more expensive than other volatiles; for economic use, it is recommended to use Desflurane with a low flow (up to 2L) anaesthetic technique.

Isoflurane is the most commonly used volatile anaesthetic agent at Dr. George Mukhari Academic Hospital. Concerns about the increased cost of desflurane compared to isoflurane limits the use of this novel agent in the public sector in South Africa. Following an extensive literature review, no studies could be found comparing quality of recovery between desflurane and isoflurane using a validated quality of recovery tool like the QoR-15.

The research question in this study is whether there is a clinically significant difference in post-operative quality of recovery (using the QoR-15 score) between desflurane and isoflurane inhalational anaesthesia in adult patients presenting for elective ophthalmological surgery under general anaesthesia.

This study will therefore compare quality of recovery between desflurane and isoflurane inhalational anaesthesia. Furthermore, the study will evaluate the relative cost of using either volatile with a basal flow anaesthetic technique.

DETAILED DESCRIPTION:
Aims & Objectives:

The aim of this study is to compare quality of recovery between desflurane and isoflurane inhalational anaesthesia. The primary objective of the study is to evaluate whether there is a difference between post-operative quality of recovery in patients who received desflurane and in patients who received isoflurane for maintenance of anaesthesia, using the QoR-15 score, a patient-rated outcome measure.

Isoflurane is the standard drug used at Dr. George Mukhari Academic Hospital theatre complex for maintenance of anaesthesia and will therefore be used as the drug for the control group. Desflurane will be used as the interventional drug. The minimal clinically important difference for the post-operative QoR-15 has been found to be 8. In other words, an intervention that changes the mean post-operative score by 8, can be interpreted to signify a clinically important improvement or deterioration.

The null hypothesis for this study is that there is no statistically significant difference in mean post-operative QoR-15 scores of patients receiving isoflurane and desflurane for maintenance of anaesthesia. The alternative hypothesis is that there is a statistically significant difference in mean post-operative QoR-15 scores between patients receiving isoflurane and desflurane.

A secondary objective will be to compare the consumption and relative cost of using isoflurane vs desflurane with a minimal or basal flow anaesthetic technique. This will be done by comparing the amount of vapour used in millilitre per hour between desflurane and isoflurane during basal flow anaesthesia. The relative cost of the vapour used will be estimated, based on the current government purchase price of isoflurane and desflurane.

Furthermore, the difference in time spent in recovery between the two patient groups will also be compared.

Methods:

This study will be conducted as a randomised, controlled, patient and observer blinded, single-centre trial with two parallel groups and a primary end-point of 15-point Quality of Recovery Score on day 1 after surgery. Randomization will be performed as block randomization with a 1:1 allocation.

The study will be conducted in the theatre complex at Dr. George Mukhari Academic Hospital, a tertiary training centre affiliated with Sefako Makgatho Health Sciences University. Specifically, the study will be conducted in the ophthalmological theatre, on patients undergoing ophthalmological surgery under general anaesthetic.

Sample size calculation is based on estimation of the difference in mean post-operative Quality of Recovery (QoR) scores, after anaesthesia with desflurane or isoflurane. With a sample size of 85 in each group, a two-sided two-sample t-test at the 5% significance level, will have 80% power to detect a difference of 8 between the mean post-operative QoR scores with desflurane and isoflurane, assuming a standard deviation of 18.5, Sample size calculation was done on nQuery Advanced (Statistical Solutions Ltd, Cork, Ireland), Release 8.0. A sample of 170, randomised in a 1:1 ratio to treatment with desflurane and isoflurane (85 per group) is proposed for this study.

Recruitment will be done by the Chief Investigator. The following steps will be followed:

1. Review the theatre booking list for theatre 11 the day before surgery.
2. Identify adult patients between the ages of 18 and 80 on the list, scheduled for general anaesthesia.
3. Review the patients in the ward:

   a. Screen for any exclusion criteria.
4. Once confirmed that there are no exclusion criteria:

   1. Explain the objectives of the study to the patient.
   2. Hand the patient a patient information leaflet and discuss any questions the patient may have.
   3. Take informed consent if the patient agrees to participate in the study.
5. Record the patient's name on a sequentially numbered list. This will be the only document to contain any personal information of the patient. It will be stored securely by the Chief Researcher. The number on the list will be the patient's study number and this number will be recorded on all study documents

Patients will be randomly allocated to either the control or the intervention group by computer randomisation. Randomisation and allocation will be managed remotely by the statistician, who will not be involved in patient care, and who will only gain access to study data after completion of data collection.

Block randomisation will be done to ensure that an equal number of patients are assigned to each treatment arm. Random block sizes will be used and the chief investigator, research assistant and treating anaesthetists will be blind to the size of each block.

Sequentially numbered, sealed, opaque envelopes will be prepared by the statistician. This will include a piece of paper indicating the group the patient has been randomised to. The sealed envelope will be handed to the treating anaesthetist on the day of surgery by the Chief Researcher. The Chief Researcher will be responsible for enrolment and assignment of participants.

The patient will be blinded to the group they have been randomised to, as the vapour will only be started after induction of anaesthesia. The research assistant administering the post-operative QoR-15 will be blinded to the intervention.

The treating anaesthetist, the Chief Researcher and theatre staff will not be blinded to the intervention, as this would not be practical. All treating anaesthetists and theatre staff will be strongly inculcated not to disclose the allocation status of the participant at any time prior or after the general anaesthetic.

The piece of paper indicating the group will be attached to the Case Report Form. The Case Report Form will be collected by the Chief Researcher and will not be in the patient's file where it may unblind the patient or research assistant.

There are no circumstances under which unblinding will be permissible.

Patients will be assessed by the chief researcher pre-operatively on the day before surgery. The demographic information on the Data Collection Form (Section A) will be completed. Information will be obtained from the patient's file, as well as from an interview with the patient. The chief researcher will accurately measure the patient's weight and height with the available scales and measuring devices in the wards.

Patients will then be asked to complete the QoR-15 in the language of their choice, as a measure of health status over the previous 24 hours. As far as possible, the QoR-15 form will be handed to the patient to complete by themselves. However, in cases where patients are visually impaired, the items on the questionnaire will be read to the patinet, and their responses recorded.

The following day, the treating anaesthetist will complete the information about the procedure in Section B of the Data Collection Form: anaesthetic time, amount of vapour used, additional medication administered, recovery time, any adverse events (bronchospasm, laryngospasm, post-operative nausea and vomiting and/or other), and whether the prescribed anaesthetic protocol was followed.

Post-operatively, a blinded observer (research assistant) will review the patient on the day following their surgery, prior to discharge. The patients will complete the QoR-15 again, as above.

As follow-up will be done before discharge, retention of patients to follow-up should not present any difficulties.

Data Management:

All study documents will be printed. All data will be recorded by hand on paper forms. After recruitment, the Chief Researcher will record the sequential study number on all documents relating to a particular patient.

The data will be captured electronically on the REDCap database by the research assistant (19). REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources.

Data from each patient will be captured on REDCap sequentially so that the study number correlates with the database entry number.

Study documents will be stored securely by the Chief Researcher. Documents will be kept in a dedicated lever-arch file and will be arranged sequentially according to study number. All study documents relating to a single patient will be stored together.

In case of incomplete data in Section B of the Data Collection Form, the chief researcher will review the following source documents in the order listed to obtain the information:

Missing data on medication given intra-operatively:

1. Blue anaesthesia report card
2. Nursing theatre record
3. Theatre record book

Missing data on medication given post-operatively:

1. Blue anaesthesia report card
2. Nursing theatre record

Missing data on anaesthesia start/end times:

1. Blue anaesthesia report card
2. Nursing theatre record
3. Anaesthetic workstation stored history
4. Theatre record book

Missing data on vapour start/end times:

1. Blue anaesthesia report card
2. Anaesthetic workstation stored history

Missing data on millilitres vapour used:

1. Anaesthetic workstation stored history

The Chief Researcher will periodically monitor the completed study documents and the database entries. If any problems are found with completion of study documents, training sessions will be arranged in the Department of Anaesthesia.

Statistical Analysis:

Demographic and clinical characteristics of patients will be summarised descriptively. Continuous variables (e.g. age or weight) will be summarised by mean, standard deviation, median, interquartile range, minimum and maximum values. Categorical variables (e.g. ethnicity or ASA status), will be summarised by frequency count and percentage calculations.

QoR scores will be considered as a continuous variable and will be summarised as above per treatment group (desflurane and isoflurane).

The null hypothesis for this study is that there is no statistically significant difference in mean post-operative QoR-15 scores of patients receiving isoflurane and desflurane for maintenance of anaesthesia. The alternative hypothesis is that there is a statistically significant difference in mean post-operative QoR-15 scores between patients receiving isoflurane and desflurane.

Based on the available literature, it is assumed that the quality of recovery scores will follow a normal distribution. The data will be inspected for normality prior to analysis.

For the primary objective, the mean and median difference in post-operative QoR-15 scores between the two groups will be tested for significance by the two-sided two-sample t-test and the nonparametric Wilcoxon rank sum test respectively. The mean and median difference between the pre-operative and post-operative QoR-15 scores for the two groups will also be tested for significance by the two-sided two-sample t-test and the nonparametric Wilcoxon rank sum test respectively.

For the secondary objectives, mean and median difference in consumption of vapour and time spent in recovery will be tested for significance by the t-test and Wilcoxon test as above.

Analysis, or comparisons, of subgroups of patients may be performed if it would be of clinical interest; for example, if there appears to be a significant difference in QoR scores between male and female patients.

Results will be presented in tables and graphs or verbatim, as applicable. All statistical analyses will be performed on SAS (SAS institute Inc, Carey, NC, USA), Release 9.4 or higher, running under Microsoft Windows for a personal computer. Statistical tests will be two-sided and p values ≤0.05 (5%) will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18-80 years of age.
* Patients presenting for ophthalmological surgery under general anaesthesia.
* ASA I and II.
* Literate in English, Setswana or Afrikaans.

Exclusion Criteria:

* Patients outside the specified age range.
* ASA III and above.
* Patients with contra-indications to Laryngeal Mask Airway use during general anaesthesia.
* Patients with severe medical or surgical conditions, who are expected to have prolonged admissions or ICU admissions.
* Patients with uncontrolled psychiatric conditions like depression, schizophrenia, mania, dementia.
* Patients with known allergy or adverse reaction to volatile anaesthetics.
* Patients with known or suspected susceptibility to Malignant Hyperthermia.
* Patients with incomplete records (Data Collection Form and QoR-15).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Post-operative Quality of Recovery score, assessed by QoR-15, change from baseline QoR-15 score pre-operatively | Pre-operative day 0 and Post-operative day 1
  A baseline 15-Item Quality of Recovery score (QoR-15) will be measured pre-operatively, and a repeat will be done on Day 1 post-operatively.
  The QoR-15 is a 15-item score evaluating both physical and mental well-being by assessing five dimensions: emotional state, physical comfort, psychological support, physical independence and pain. Each of the 15 items are scored by the patient from 0 (worst score) to 10 (best score), giving a lowest possible score of 0 (worst outcome), and a highest possible score of 150 (best outcome). This continuous composite score allows comparisons between intervention groups. The minimal clinically important difference (MCID) and patient acceptable symptom state score for the QoR-15 score has been determined: the MCID is 8 and the acceptable symptom state score is 118.

SECONDARY OUTCOMES:
Consumption of anaesthetic vapour with basal anaesthetic technique | Intraoperative day 0
  The vapour use per case in millilitres of isoflurane or desflurane will be recorded from the anaesthetic machine.
Cost of anaesthetic vapour with basal to minimal flow anaesthetic technique | Intraoperative day 0
  Calculating cost of isoflurane and desflurane used based on consumption and cost data from hospital pharmacy.
Time spent in post-operative recovery unit | Post-operative day 0
  The time the patient enters and leaves the post-operative recovery room will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Charlé Steyl, MBChB DA FCA, Principal Investigator — Sefako Makgatho Health Sciences University
Locations (1):
- Sefako Makgatho Health Sciences University, Ga-Rankuwa, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Anonimized data will be made available in appendices/supplements to the final publication, for other researchers to review results, or to include in systematic reviews/meta-analyses. All IPD that underlie results in the publication will be made available, but no personal information of patients will be released.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be available after writing up the study, it will be included in the MMed thesis as well as in appendices/supplements to final publication. The IPD will be available indefinitely.
Access Criteria: Anyone who accesses the final publication will be able to review the anonimized IPD through the appendices/supplements to the final publication.

REFERENCES:
- [Derived] Steyl C, Kluyts HL. A randomised controlled trial comparing quality of recovery between desflurane and isoflurane inhalation anaesthesia in patients undergoing ophthalmological surgery at a tertiary hospital in South Africa (DIQoR trial). BJA Open. 2023 Dec 20;9:100246. doi: 10.1016/j.bjao.2023.100246. eCollection 2024 Mar. PMID 38193018

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT04188314/Prot_SAP_ICF_002.pdf